CLINICAL TRIAL: NCT05031247
Title: Mental Health and Wellness Pilot Study Among Aging Immigrants and Refugees
Brief Title: Refugee Mental Health and Wellness Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Hafifa Siddiq, PhD, RN, MSN, Postdoctoral Fellow, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-000174
Record Dates: First submitted 2021-06-11; First posted 2021-09-01 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Social Isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Navigator Social Support (Experimental): More intensive case management and weekly check-ins with older adults. The Community Navigator will be focused on increasing social contact and connection for older adult refugees and immigrants. Those who receive the intervention will be offered up to ten (30-minute-long) meetings with a Community Navigator and access to up to three group sessions over a 3-month period, alongside the standard services they receive for enrollment with the organization.
  Interventions: Other: Wellbeing Program
- Program Support as Usual (No Intervention): Standard program support will be provided to participants enrolled. These services are offered to all enrolled in the program and may include, but is not limited to the following: financial assistance services, case management, healthcare access services, employment and tax services, education services, citizenship and immigration services, community services and civic engagement, and refugee services.

INTERVENTIONS:
Other: Wellbeing Program — The community navigator program was developed during a three-phase community-based participatory research project that aims to examine emotional/mental health needs and address access to mental health services among immigrants and refugees from Muslim-majority countries.
  Other Names: Community Navigator
  Arms: Community Navigator Social Support

SUMMARY:
This pilot study will develop and examine the acceptability of a Community Navigator program of support for 10-24 older adult Arab Americans participants receiving services at a refugee-serving organization based in Southern California. This program will provide participants with social support from a 'Community Navigator,' who will work with clients to help promote attendance and engagement with the community during social activities and community events. This program aims to reduce feelings of loneliness or social isolation. In partnership with the refugee-serving organization, the UCLA investigators will implement this program in addition to services provided as usual at the community partner site. Researchers will then conduct interviews to explore participants' experiences and perceptions for improvement of the program.

DETAILED DESCRIPTION:
The Refugee Mental Health and Wellness Pilot Study aims to increase community connections and reduce loneliness for older adult immigrants and refugees, specifically from MENA countries of origin through the implementation of a Community Navigator program. This program will be implemented within an existing aging program for older adults at a refugee-serving organization that provides social services, English language classes, and computer classes for this population. The pilot program is an extension of case management services at this organization. The program provides up to ten weekly virtual (through video or telephone) home-visiting sessions. During these sessions, an Arabic-speaking program coordinator or an Arabic-speaking nurse will assess client wellbeing, social service needs, as well as referral to social activities and other services needed over three months. The coordinator or nurse will be trained in a trauma-informed approach to working with refugee and immigrant clients. Participants will be recruited at the partner site. This study aims to recruit between 10-24 older adults interested in participating in semi-structured interviews to examine program acceptability and explore suggestions on improving the program. The baseline and completion survey will collect data on social demographics, social support, depressive symptoms, and loneliness score. Interviews will be conducted at least 6-8 weeks upon enrollment in the program. This pilot study will provide preliminary evidence of the acceptability of Community Navigator support and trial evaluation procedures for testing this. The results will inform a future feasibility study and potentially, and potentially, a randomized controlled trial of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults who self-identify as Arab or Middle Eastern/North Africa over the age of 55

Exclusion Criteria:

* For all participants, those who do not have the capacity to consent to participate.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Revised UCLA Loneliness Scale (R-UCLA) | 12 weeks
  Decreased loneliness will be measured using the Revised UCLA Loneliness Scale (R-UCLA). This scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation.

SECONDARY OUTCOMES:
Lubben Social Support Network Scale | 12 weeks
  Perceived social support will be measured using the Lubben Social Support Network scale. The Lubben Social Network Scale is a six-item self-report measure assessing quantity and quality of contact with family and friends.

OTHER OUTCOMES:
Patient Health Questionnaire-9 Item Depression Scale | 12 weeks
  Depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9). The PHQ9 is a nine-item self-report measure of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hafifa Siddiq, PhD, Principal Investigator — UCLA and Charles R. Drew University

IPD SHARING:
Plan to Share IPD: No
Due to the small participant sample size and vulnerable population (older adult refugees) and risk for exposing personally identifiable information within qualitative interview data, IPD will not be shared with other researchers outside the research team.